CLINICAL TRIAL: NCT07313202
Title: Ivarmacitinib in Advanced Solid Tumors: A Prospective, Two-Cohort, Two-Phase Exploratory Study in Patients Discontinued Due to Immune Intolerance
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA-SOLID-II-004
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Patients With Advanced Solid Tumors Who Discontinued Treatment Due to irAE
MeSH Terms: interventions — ivarmacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group 1：Subjects who developed resistance or dependence to hormone therapy (Experimental)
  Interventions: Drug: Ivarmacitinib
- Treatment group 2：Subjects whose irAE has resolved to Grade ≤1 (Experimental)
  Interventions: Drug: Ivarmacitinib

INTERVENTIONS:
Drug: Ivarmacitinib — 8 mg, orally, once daily. Cohort 1: Continue dosing until irAE resolves to ≤ Grade 1, with a maximum treatment duration of 28 days.
  Arms: Treatment group 1：Subjects who developed resistance or dependence to hormone therapy
Drug: Ivarmacitinib — Cohort 2: Combination therapy with ICIs, with a maximum treatment duration not exceeding the duration of ICI administration.
  Arms: Treatment group 2：Subjects whose irAE has resolved to Grade ≤1

SUMMARY:
This study is a Phase II, two-cohort, multicenter, two-stage clinical trial. It plans to enroll 72 subjects with solid tumors who discontinued prior ICI therapy due to irAE. Cohort 1 enrolls subjects with irAE resistant to or dependent on corticosteroid therapy. Subjects in Cohort 1 who achieve ≤ Grade 1 irAE resolution following treatment may then enroll in Cohort 2. Cohort 2 enrolls subjects with irAE achieving ≤ Grade 1 resolution following treatment, and deemed eligible for ICI re-initiation by the investigator. Phase I is the safety run-in phase, enrolling 6 subjects per cohort. Phase II is the expansion phase, enrolling 30 subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. ECOG performance status score 0-1.
3. Expected survival ≥ 12 weeks.
4. Solid tumor patients who have discontinued treatment with immune checkpoint inhibitors (ICIs).
5. Treatment with ICIs may be administered as monotherapy or in combination with other therapies (including but not limited to radiotherapy, chemotherapy, targeted therapy, etc.).
6. Current Status of irAE:

   Cohort I:
   1. Patients currently diagnosed with steroid-resistant or steroid-dependent immune-related adverse events (immune myocarditis, immune colitis, immune myositis-arthritis, immune skin reactions, immune hepatitis, etc.);
   2. Patients with contraindications to steroid use, or who refuse continued steroid therapy due to adverse reactions following steroid administration.

   Cohort II:
   1. Patients discontinued immunotherapy due to irAE (CTCAE 5.0) after receiving ≥1 line of treatment including ICIs;
   2. Time since discontinuation of immunotherapy due to irAE ≤3 months;
   3. irAE has resolved to ≤Grade 1.
7. The patient still possesses certain organ and bone marrow functions:

   Cohort 1:
   1. Hemoglobin ≥90 g/L, neutrophil count ≥1.0 × 10^9/L, platelet count ≥75 × 10^9/L; lymphocyte count ≥0.5 × 10^9/L; coagulation function: INR, APTT, and PT all ≤1.5 × UNL;
   2. Liver function: Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 3 × ULN, alanine aminotransferase (ALT) ≤ 3 × ULN. For patients with immune hepatitis, specific liver function biochemical parameters are not restricted; adequate liver function is defined as Child-Pugh class A-B;
   3. Renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min;
   4. Or patients assessed by the investigator as having adequate organ function.

   Cohort II:

   Organ function levels must meet the following requirements (no blood transfusion or hematopoietic growth factor therapy within 2 weeks prior to blood screening):
   1. ANC ≥ 1.5 × 10⁹/L;
   2. PLT ≥ 100 × 10⁹/L;
   3. Hb ≥ 90 g/L;
   4. TBIL ≤ 1.0 × ULN;
   5. ALT and AST ≤ 2.5 × ULN;
   6. BUN and Cr ≤ 1.5 × ULN.
8. All women of childbearing potential must have a negative serum pregnancy test during the screening period and must use reliable contraception from signing the informed consent form until 3 months after the last dose.
9. Subjects voluntarily participate in this study, sign the informed consent form prior to the screening process, demonstrate good compliance, and cooperate with safety follow-up.
10. The subject is judged by the investigator to be able to adhere to the study protocol.

Exclusion Criteria:

* 1) Individuals with allergic diseases, a history of severe drug allergies, or potential hypersensitivity to Ivarmacitinib or its components; 2) Patients diagnosed with an embolic event within 3 months prior to enrollment, excluding superficial venous thrombosis (e.g., deep vein thrombosis, pulmonary embolism, embolic stroke, myocardial infarction, or peripheral arterial insufficiency); 3) Patients with severe non-irAE-related cardiac, hepatic, renal, or systemic diseases; 4) Patients with active tuberculosis or who received live vaccines during the illness period; 5) Patients with uncontrolled infectious diseases; 6) Patients with moderate to severe heart failure (NYHA Class III/IV); 7) Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) positive, with hepatitis B virus (HBV) deoxyribonucleic acid (DNA) exceeding 500 IU/mL or 1000 copies per milliliter (cps/mL); Hepatitis C virus (HCV) antibody (HCV-Ab) positive with HCV RNA quantitative levels exceeding the upper limit of normal for the assay; HIV antibody (Anti-HIV) positive; active syphilis. Meeting any one of the above criteria.

  8) Previous treatment with JAK inhibitors prior to enrollment (for Cohort 1: ≤30 days of prior JAK inhibitor use, irAE resolution ≤ Grade 1, and investigator assessment permitting ICI restart; eligible for Cohort 2); 9) Cohort 2 participants with prior ICI restart therapy, including but not limited to PD-1/PD-L1 inhibitors, CTLA-4 inhibitors, etc.; 10) Patients receiving intravenous biologic therapy for other baseline autoimmune diseases; 11) Pregnant or lactating females, and males or females unwilling to use contraception; 12) Psychiatric disorders impairing study compliance; 13) Subjects deemed unsuitable for this study by the investigator shall be excluded, such as those judged to have other factors that may necessitate premature termination of the study. These include: - Concurrent treatment for other serious illnesses (including psychiatric disorders) - Severe laboratory abnormalities - Family or social circumstances that may compromise subject safety or interfere with data/sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-26 (Estimated)

PRIMARY OUTCOMES:
Response rate to adverse reactions during the treatment cycle | In the study, treatment was administered on day 30 after the last dose.
Discontinuation rate due to irAE | Follow-up visits were conducted every 30 days from the last dose of treatment until 90 days.

IPD SHARING:
Plan to Share IPD: No